CLINICAL TRIAL: NCT06081894
Title: A Phase 3, Multi-Center, Randomized, Double-Blind Trial to Evaluate the Efficacy and Safety of Aficamten Compared to Placebo in Adults With Symptomatic Non-Obstructive Hypertrophic Cardiomyopathy
Brief Title: Phase 3 Trial to Evaluate the Efficacy and Safety of Aficamten Compared to Placebo in Adults With Symptomatic nHCM
Acronym: ACACIA-HCM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Collaborators: Sanofi (Industry); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CY 6033; 2023-505797-15-00 (Other: EU CTR Number)
Record Dates: First submitted 2023-08-31; First posted 2023-10-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Symptomatic Non-Obstructive Hypertrophic Cardiomyopathy
Keywords: CK-3773274; CK-274; Aficamten; Symptomatic Non-Obstructive Hypertrophic Cardiomyopathy; nHCM; ACACIA-HCM; ACACIA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aficamten (Experimental): Participants in this arm will receive a single daily oral dose of 5 mg, 10 mg, 15 mg, or 20 mg of aficamten with dose levels guided by echocardiography assessments, for up to 72 weeks.
  Interventions: Drug: Aficamten
- Placebo (Placebo Comparator): Participants in this arm will receive placebo, for up to 72 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aficamten — Oral Tablet
  Arms: Aficamten
Drug: Placebo — Oral Tablet
  Arms: Placebo

SUMMARY:
This clinical trial will study the effects of aficamten (versus placebo) on the quality of life, exercise capacity, and clinical outcomes of patients with non-obstructive hypertrophic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-85 years of age
* Body mass index < 40 kg/m2
* Diagnosed with nHCM and has a screening echocardiogram with the following:

  * End-diastolic left ventricular (LV) wall thickness:

    * ≥ 15 mm in one or more myocardial segments OR
    * ≥ 13 mm in one or more wall segments and a known disease-causing gene mutation or positive family history of HCM AND
    * Resting LVOT-G < 30 mmHg AND Valsalva LVOT-G < 50 mmHg AND
    * LVEF ≥ 60%
  * Participants with a history of intracavitary obstruction are eligible.
* NYHA class II or III
* Respiratory exchange ratio of ≥ 1.00 at screening by cardiopulmonary exercise testing (CPET) and predicted peak oxygen uptake (pVO2) ≤ 90% for age and sex
* KCCQ-CSS score of ≤ 85
* NT-proBNP of:

  * NT-pro BNP ≥ 300 pg/mL or NT-proBNP ≥ 900 pg/mL if in atrial fibrillation or atrial flutter OR
  * For Black participants, an NT-pro BNP ≥ 225 pg/mL or NT-proBNP ≥ 675 pg/mL if in atrial fibrillation or atrial flutter

Exclusion Criteria:

* Significant valvular heart disease (per Investigator judgment)

  * Moderate or severe valvular aortic stenosis or fixed subaortic obstruction
  * Moderate or severe mitral regurgitation
* Known or suspected infiltrative, genetic or storage disorder causing cardiac hypertrophy that mimics nHCM (eg, Noonan syndrome, Fabry disease, amyloidosis)
* Known current unrevascularized coronary artery stenosis of ≥ 70% or documented history of myocardial infarction.
* History of LV systolic dysfunction (LVEF < 45%) or stress cardiomyopathy
* Inability to exercise on a treadmill or bicycle (eg, orthopedic limitations)
* Documented room air oxygen saturation reading < 90% at screening or history of significant chronic obstructive pulmonary disease or severe/significant pulmonary hypertension
* History of syncope, symptomatic ventricular arrhythmia, or sustained ventricular tachyarrhythmia with exercise within 3 months prior to screening
* History of resistant hypertension (persistently elevated blood pressure despite maximal doses of 3 or more classes of medications for hypertension control)
* Screening diastolic blood pressure ≥ 100 mmHg
* Received prior treatment with aficamten
* Received treatment with mavacamten within 3 months prior to screening (must be discussed with the medical monitor prior to screening)
* Undergone septal reduction therapy < 6 months prior to screening
* Is being considered for or is likely to be considered for heart transplant listing or left ventricular assist device placement during the study period
* Paroxysmal or permanent atrial fibrillation is excluded only if:

  * rhythm restoring treatment (e.g., direct-current cardioversion, atrial fibrillation ablation procedure, or antiarrhythmic therapy) has been required ≤ 3 months prior to screening
  * rate control and anticoagulation have not been achieved for at least 3 months prior to screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Kansas City Cardiomyopathy Questionnaire - Clinical Summary Score (KCCQ-CSS) | Baseline to Week 36
  Effect of aficamten compared with placebo on participant health status
Change in pVO2 | Baseline to Week 36
  Effect of aficamten compared with placebo on maximal exercise capacity

SECONDARY OUTCOMES:
Change in composite of two Z-scores of CPET parameters (pVO2 and VE/VCO2 slope) | Baseline to Week 36
  Effect of aficamten compared with placebo on global exercise capacity based on maximal and sub-maximal exercise performance
Proportion of participants with ≥ 1 class improvement in NYHA Functional Class | Baseline to Week 36
  Effect of aficamten compared with placebo on NYHA Functional Classification
Change in NT-proBNP | Baseline to Week 36
  Effect of aficamten compared with placebo on a biomarker of cardiac wall stress
Change in LAVI in participants without atrial fibrillation or flutter at baseline on ECG | Baseline to Week 36
  Effect of aficamten compared with placebo on echocardiographic measures of structural remodeling
Time to first CV event | Baseline to End of Study, Week 72
  Effect of aficamten compared with placebo on cardiovascular events (ie, CV death, heart transplantation or left ventricular assist device, aborted sudden cardiac death, non-fatal stroke, heart failure hospitalization, or cardiac arrhythmia (atrial fibrillation or ventricular tachyarrhythmia) requiring treatment or hospitalization)

CONTACTS AND LOCATIONS:
Overall Officials: Cytokinetics MD, Study Director — Cytokinetics
Locations (180):
- United States (60):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC San Diego Health - Sulpizio Cardiovascular Center, La Jolla, California
  - Keck Medical Center of USC (Outpatient Clinic), Los Angeles, California
  - Cedars-Sinai Medical Center (Smidt Heart Institute), Los Angeles, California
  - UCLA Medical Center Cardiovascular Clinic, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Medical Group - Cardiology Associates, Fort Lauderdale, Florida
  - Investigational Drug Services, AdventHealth Orlando, Orlando, Florida
  - Emory Clinic, Atlanta, Georgia
  - Piedmont Heart Institute (CPET), Fayetteville, Georgia
  - The Queen's Medical Center-Punchbowl, Honolulu, Hawaii
  - Northwestern University, Evanston, Illinois
  - Ascension St. Vincent, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - M Health Fairview University of Minnesota Medical Center - East Bank, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Northwell Health North Shore University Hospital, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Sanger Heart & Vascular Institute - HCM Clinic, Charlotte, North Carolina
  - The Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Ascension Saint Thomas Heart West, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Health, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Health Care Services, Falls Church, Virginia
  - VCU Health Downtown Medical Campus, Richmond, Virginia
  - Carilion Clinic Cardiology, Roanoke, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Providence Sacred Heart Medical Center & Children's Hospital (CPET), Spokane, Washington
  - WVU Medicine, Morgantown, West Virginia
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Italiano de Buenos Aires Juan Domingo Peron, Buenos Aires
  - ICBA - Instituto Cardiovascular de Buenos Aires, Buenos Aires
  - Hospital Privado Centro Medico de Cordoba S.A, Córdoba
- Australia (3):
  - The Prince Charles Hospital, Chermside, Queensland
  - Flinders Medical Centre Cardiology Research, Adelaide, South Australia
  - Fiona Stanley Hospital, AHF Unit, Murdoch
- Brazil (9):
  - Instituto D'Or de Pesquisa e Ensino/Cardio Pulmonar da Bahia SA, Ondina, Salvador
  - Fundacao Felice Rocho / Hospital Felicio Rocho, Minas Gerais
  - NUPEC Cardio / Cardio HVC, Minas Gerais
  - CLINICOR Clinica Cardiologica LTDA, Ribeirão Preto
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Instituto do Coracao do Hospital de Aguiar, São Paulo
  - Associacao Lar Sao Francisco de Assis na Providencia de Deus - Hospital Universitario Sao Francisco na Providencia de Deus (HUSF), São Paulo
  - Saraiva & Berlinger LTDA - EPP/IPECC - Instituto de Pesquisa Clinical de Campinas, São Paulo
  - Hospital das Clinicas de Faculdade de Medicina de Ribeirao Preto da Universidade de Sao Paulo - HCFMRP, São Paulo
- Canada (5):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Health Sciences North, Greater Sudbury, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - QEII Health Science Centre (Halifax Infirmary site), Halifax
- China (12):
  - The 1st Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Peking University First Hospital, Beijing
  - Fuwai Hospital, CAMS & PUMC, Beijing
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Hospital of Jilin University, Jilin
  - Zhongda Hospital Southeast University, Nanjin
  - Shanghai Ruijin Hospital Luwan Branch, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - People's Hospital of Liaoning Province, Shenyang
  - Remin Hospital of Wuhan University, Wuhan
  - The 1st affi. Hospital of Xi'an Jiaotong University, Xi'an
  - The 1st affiliated Hospital of Zhengzhou University, Zhenzhou
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Department of Cardiology Copenhagen University Hospital, Bispebjerg, Copenhagen
  - Odense University Hospital, Department of Cardiology, Odense
- France (8):
  - Assistance Publique Hopitaux de Marseille, Marseille
  - Clinique Du Millenaire, Montpellier
  - Centre Hospitalier Universitaire De Montpellier, Montpellier
  - Assistance Publique Hopitaux De Paris, Paris
  - Assistance Publique Hopitaux de Paris, Paris
  - Centre Hospitalier Universitaire De Bordeaux, Pessac
  - Centre Hospitalier Universitaire De Nantes, Saint-Herblain
  - Hopital Rangueil, Toulouse
- Germany (4):
  - Charite-Universitaetsmedizin Berlin Campus Virchow-Klinikum (CVK) Medizinische Klinik mit Schwerpunkt Kardiologie, Berlin
  - Herzzentrum der Universitatsmedizin Gottingen, Göttingen
  - Universitaesklinkum Heidelberg Klinik fuer Kardiologie, Angeiologie und Pneumologie, Heidelberg
  - Univeristy Hospital Jena Clinic for Internal Medicine I (Cardiology, Angiology, Internal Intensive Care Medicine), Jena
- Greece (4):
  - Evangelismos General Hospital of Athens, Athens
  - "Hippokration" General Hospital of Athens, Athens
  - University General Hospital Attikon, Attiki
  - Onassis Cardiac Surgery Center, Kallithea
- Hungary (2):
  - Semmelweis Egyetem Varosmajori Sziv- es Ergyogyaszati Klinika, Budapest
  - University of Szeged, Szeged
- Landspitali University Hospital, Reykjavik, Iceland
- Israel (5):
  - The Barzilai University Medical Center 2 - Cardiology Division, Ashkelon
  - Division of Cardiology Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - The Chaim Sheba Medical Center, Ramat Gan
  - Ziv Medical Center, Safed
- Italy (10):
  - Cardiology Department IRCCS San Donato Hospital - University of Milan, San Donato Milanese, Milano
  - UOC Cardiologica, Brescia
  - Azienda Ospedaliera Universitaria Careggi pad. 13 Clinica Medica II Plano Cardiologia, Florence
  - Cardiologia Universitaria - UTIC - Riabilitazione Cardiologica Azienda Ospedaliero Universitaria - Ospedali Riuniti, Foggia
  - Unita Operativa di Riabilitazione Cardiologica, Istituto Auxologico Italiano, IRCCS - Auxologico San Luca, Piazzale Brescia, 20, Milan
  - Dipartimento Cardio-toraco- vascolare, ASST Grande Ospedale Metropolitano, NiguardaPiazza Ospedale Maggiore, 3, Milan
  - Dipartimento di Emergenze Cardiovascolari, Medicina Clinica e dell'Invecchiamento, AOU Federico II, Napoli
  - Fondazione Toscana Gabriele Monasterio Per La ricerca Medica e Di Sanita Pubbliga (FTGM) Cardio-Toracic-UOC Cardiology and Cardiovasulcar Medicine San Cataldo Hospital at CNR, Pisa
  - Dipartimento Cardiopolmonare, Istituto di Ricovero e Cura a Carattere Scientifico San Raffaele, Roma
  - Azienda Sanitaria Universitaria Giuliano Isontina Trieste SC Cardiologia, Trieste
- Japan (22):
  - Kyushu University Hospital, Fukuoka
  - Kobe City Medical Center General Hospital, Hyōgo
  - Hyogo Prefectural Harima-Himeii General Medical Center, Hyōgo
  - University of Tsukuba Hospital, Ibaraki
  - SHOWA Medical University Fujigaoka Hospital, Kanagawa
  - Kochi Medical School Hospital, Kochi
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Mie University Hospital, Mie
  - National University Corporation Tohoku University Tohoku University Hospital, Miyagi
  - Shinshu University Hospital, Nagano
  - Osaka Metropolitan University Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - National Cerebral and Cardiovascular Center, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Osaka
  - Kitasato University Hospital, Sagamihara
  - Saitama Medical University International Medical Center, Saitama
  - Hamamatsu University Hospital, Shizuoka
  - St. Luke's International Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
  - Teikyo University Hospital, Tokyo
- Netherlands (3):
  - P. Debyelaan 25, Maastricht, HX
  - Amsterdam UMC, location AMC, Amsterdam
  - Erasmus University Medical Center, Rotterdam
- Kardio Brynow Sp. z o.o., Katowice, Poland
- Portugal (5):
  - Unidade Local de Saude do Alto Ave, E.P.E, Creixomil, Guimaraes
  - Unidade Local de Saude da Regiao de Aveiro, E.P.E., Aveiro
  - Unidade Local de Saude de Sao Jose, E.P.E, - Hospital de Santa Marta Servico de Cardiologia, Lisbon
  - Hospital da Luz, Lisbon
  - Hospital CUF Descobertas, Lisbon, Cadiology Department, Lisbon
- Spain (13):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón (HGUGM), Calle del Doctor Esquerdo, 46., Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Virgen de la Victoria Campus Universitario de Teatinos, Málaga
  - Hospital Clinico Universitario Virgen de la, Murcia
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Alvaro Cunqueiro, Vigo
- United Kingdom (7):
  - NHS Tayside Ninewells Hospital & Medical School, Dundee, Scotland
  - NHS Greater Glasgow and Clyde Queen Elizabeth University Hospital, Glasgow
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust St Bartholomew's Hospital, London
  - St George's University Hospitals NHS Foundation Trust,, London
  - Royal Brompton Hospital, London
  - Oxford Centre for Clinical Magnetic Resonance Research (Ocmr), Oxford

IPD SHARING:
Plan to Share IPD: No